CLINICAL TRIAL: NCT01672710
Title: Pilot Study of Application of the Hubbard Detoxification Program to Veterans With Gulf War Illness
Brief Title: Gulf War Illness: Evaluation of an Innovative Detoxification Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University at Albany (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The Sage Colleges (Other); Women's College Hospital (Other); Severna Park Health and Wellness Center (Unknown)
Responsible Party: Principal Investigator, David O. Carpenter, Director, Institute for Health and the Environment, University at Albany, University at Albany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GW093066
Record Dates: First submitted 2012-08-15; First posted 2012-08-27 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Gulf War Illness
Keywords: Hubbard detoxification; Exercise; Sauna therapy; Niacin; Gulf War illness
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Steam Bath

STUDY DESIGN:
Intervention Model Description: Pilot
Oversight: Data Monitoring Committee: No

ARMS (2):
- regimen of niacin, exercise, sauna, (Experimental): 4-5 week daily sauna, exercise and niacin with other supplements
  Interventions: Drug: plain crystalline niacin, exercise, sauna
- waitlist (Other): 4 week waitlist with treatment as usual
  Interventions: Drug: plain crystalline niacin, exercise, sauna

INTERVENTIONS:
Drug: plain crystalline niacin, exercise, sauna — A four to six week regimen consisting of daily, supervised, mild-moderate exercise as tolerated for 20 minutes, supervised, intermittent Finnish saunas (at about 140'F) sauna time with breaks and showers, gradually increased as tolerated to approximately 4 hours, dietary supplements including immediate release niacin in gradually increasing doses from 100 mg to a maximum of 5000 mg per day, salt and water, other vitamins, minerals and oils per Hubbard protocol.
  Other Names: Hubbard detoxification program

SUMMARY:
Gulf War illness is found in about one fourth of veterans of the 1990-1991 Gulf War and is characterized by persistent memory and concentration problems, headaches, fatigue and muscle and joint pain. It is not known what causes the illness, but exposure to chemicals is suspected. The Hubbard detoxification program consists of exercise and sauna therapy together with administration of several dietary supplements, particularly crystalline niacin used at increasing concentrations over a period of about four weeks. The investigators hypothesize that this program will reduce symptoms, as tested by administration of cognitive and quality of life tests and serum clinical chemistry tests.

DETAILED DESCRIPTION:
This will be a pilot randomized controlled trial of feasibility, safety and changes in fatigue and pain symptoms, measured quality of life, mental health status, and neuro-cognitive functioning of a group of GWVs after a 4 to 6 week sauna detoxification regimen as compared to control. For control subjects we will also have a group of GWVs receiving usual care who are randomly assigned to a waitlist and who will start the intervention after a four to six week delay. The waitlist group will also take part in the baseline tests a second time just prior to their treatment 4 to 6 weeks later and a 7-day post-treatment battery of tests the same as described for the treatment group. Finally, there will be a 3-month follow-up with both the groups. The Severna Park Health and Wellness Center (SPHWC) is a commercial center that offers the Hubbard detoxification program. The investigators will contract with SPHWC to provide the program to the subjects of this study and to provide office space for the Study Coordinator, so that all components of this project except the initial Physician evaluation and blood sample acquisition can be done at the Center, not just the detoxification.

Study Variables: The investigators will examine feasibility of the research design, and safety of the regimen and estimate changes in:

* Quality of life as measured by the Veterans Short Form (SF36-V). The SF36-V also includes physical (PCS) and mental (MCS) component summary scores.
* Case status for GWI will be assessed utilizing the Kansas criteria.
* Symptoms of fatigue and pain in GWI will be measured wit, the Multidimensional Fatigue Inventory, and the short-form McGill Pain-2 Questionnaire.
* Cognitive function will be measured with a battery of neurocognitive tests. These will include visual motor, memory and executive functioning as measured by the Trailmaking test, Grooved Pegboard, Wechsler Memory Abbreviated test, and the Stroop color word test. To account for potential confounding in neurocognitive testing, mental health status will be evaluated using the Symptom Checklist 90 revised and the State Trait Anxiety Inventory.
* Physical health status will be assessed via standard medical examination and laboratory analyses of serum metabolic panel, lipid profile and hormones.

Sampling Method: This will be a convenience sample and will consist of Gulf War Veterans who meet the Kansas case definition for Gulf War illness and reside in the Washington/Baltimore area or can travel to and reside in the area for several weeks. The individuals who show interest in this study, who meet eligibility criteria and subsequently agree to participate will be selected to enroll in the study.

Randomization: Volunteers will be randomly assigned to a group when they enroll. One group will be the immediate experimental intervention group and one group will be the wait-list control group. Random assignment will be achieved by use of sequentially numbered, opaque, sealed envelopes. Both will undergo the detoxification protocol, but the control group will be tested twice prior to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any veteran of the 1990-1991 Gulf War who meets the Kansas Gulf War Illness case definition.

Exclusion Criteria:

* Veterans who meet the inclusion criteria but have been diagnosed by a physician with (1) chronic conditions (eg., cancer, heart disease, diabetes, liver disease, multiple sclerosis, etc.) that are not associated with Gulf War service but can produce diverse symptoms similar to Gulf War Illness; (2) conditions that might interfere with respondents' ability to report symptoms (eg., psychiatric conditions or history of hospitalization for depression, alcohol or drug dependence; (3) pregnancy or unwillingness to use contraception.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Carpenter, MD, Principal Investigator — University at Albany
Locations (1):
- Severna Park Health and Wellness Center, Annapolis, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Graves DF, Morse GS, Kerr K, Carpenter DO. A Pilot Study to Examine Psychological and Neuropsychological Outcomes and a Novel Detoxification Program for Gulf War Illness. Mil Med. 2021 Jan 25;186(Suppl 1):205-213. doi: 10.1093/milmed/usaa486. PMID 33499551

RESULTS

PARTICIPANT FLOW:
Groups:
- Niacin, Exercise, Sauna,: plain crystalline niacin, exercise, sauna: A four to six week regimen consisting of daily, supervised, mild-moderate exercise as tolerated for 20 minutes, supervised, intermittent Finnish saunas (at about 140'F) sauna time with breaks and showers, gradually increased as tolerated to approximately 4 hours, dietary supplements including immediate release niacin in gradually increasing doses from 100 mg to a maximum of 5000 mg per day, salt and water, other vitamins, minerals and oils per Hubbard protocol.
- no Intervention: waitlisted group receives treatment as usual for 4 weeks
Period: Controlled Comparison 5 Week Follow-up
Arm/Group | Niacin, Exercise, Sauna, | no Intervention
Started | 22 | 10
Completed | 22 (sauna intervention group repeat all assessments 7 days after complete the regimen) | 10 (waitlist group repeat baseline assessments after 4 week time period then begin sauna)
Not Completed | 0 | 0
Period: Waitlist Assessed After Sauna Regimen
Arm/Group | Niacin, Exercise, Sauna, | no Intervention
Started | 22 (immediate start group no further assessments until 3 month follow up) | 10 (waitlisted group receive the 4 week intervention and complete 7 day assessments)
Completed | 22 (non applicable, cannot compare the immediate start and waitlist in this period) | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: 3 Month Follow up
Arm/Group | Niacin, Exercise, Sauna, | no Intervention
Started | 22 | 9
Completed | 16 | 5
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — follow up due after termination date | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- no Intervention: treatment as usual for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Niacin, Exercise, Sauna, | no Intervention | Total
Number analyzed (Participants) | 22 | 10 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — in years
  years | 51.7 (7.9) | 50.2 (5.5) | 51.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Short Form-36 for Veterans Quality of Life Physical Component Summary Scores
Description: Qualify of life will be determined per Short Form-36 for veterans quality of life Physical component (PCS) summary scales, range from 0 to 100 with 100 being better; 50 is expected population average.
  immediate intervention and waitlist groups changes compared from baseline and adjusted mean differences at end of 5 weeks.
Time Frame: baseline, 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Niacin, Exercise, Sauna, | no Intervention
Number analyzed (Participants) | 22 | 10
score on a scale
  baseline PCS score | 30.3 (8.9) | 36.7 (10.5)
  5 week PCS scores | 38.2 (10.3) | 35.7 (12.1)
Statistical Analysis 1: Comparison: Niacin, Exercise, Sauna, vs no Intervention; Test type: Superiority; p < 0.05, ANCOVA; Mean Difference (Net) = 6.9, 95% CI 2-sided [-0.3 to 14.2]

2. Secondary Outcome: Fatigue Severity
Description: Multidimensional fatigue inventory. change in Self reported fatigue severity. Measures 5 dimensions of fatigue: general, physical, mental, reduced motivation and reduced activity. Scores 4-20 in each dimension, higher score worse fatigue.
Time Frame: baseline, 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Niacin, Exercise, Sauna, | no Intervention
Number analyzed (Participants) | 22 | 10
score on a scale
  Baseline fatigue score | 17.4 (2.6) | 15.3 (5.3)
  5 week fatigue score | 12.8 (4.8) | 15.7 (3.6)

ADVERSE EVENTS:
Time Frame: 4-6 weeks
Groups:
- Niacin, Exercise, Sauna: the immediate intervention group (n=22) completed the step in 4 weeks,
- no Intervention Waitlist: received only usual care, followed by (n=10) crossed over to receive the intervention for a 4 week period
Arm/Group | Niacin, Exercise, Sauna | no Intervention Waitlist
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/10
Other Adverse Events (participants affected / at risk) | 3/22 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin, Exercise, Sauna (N=22) | no Intervention Waitlist (N=10)
hypotension (Cardiac disorders) | 2 (2) | NA
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No